CLINICAL TRIAL: NCT00953004
Title: Effect of Flaxseed and Flaxseed Mucilage on Energy Digestibility, Lipid Profile and Appetite
Brief Title: Flax Mucilage and Apparent Nutrient Digestibility
Acronym: HØRFRØ
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Copenhagen (Other)
Responsible Party: Head and professor Arne Astrup, University of Copenhagen, Department of Human Nutrition
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B245
Record Dates: First submitted 2009-07-17; First posted 2009-08-06 (Estimated); Last update posted 2010-11-11 (Estimated); Status verified 2009-08

CONDITIONS: Obesity
Keywords: dietary fiber; obesity; apparent energy digestibility
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- fiber drink (Experimental)
  Interventions: Dietary Supplement: fiber drink and fiber bread
- fiber bread (Experimental)
  Interventions: Dietary Supplement: fiber drink and fiber bread
- placebo (Experimental)
  Interventions: Dietary Supplement: fiber drink and fiber bread

INTERVENTIONS:
Dietary Supplement: fiber drink and fiber bread — fiber drink or fiber bread three times daily

SUMMARY:
The aim is to study the effects of flaxseed mucilage, rich in dietary fiber on apparent fat and energy digestibility in young adults.

DETAILED DESCRIPTION:
A 3 times 1-wk randomised crossover dietary intervention study, where the full diet is provided to 17 young subjects along with different flaxseed mucilage preparations. During the last five days, fecal samples are collected. Fasting blood samples are collected on day 1 and 8 in each period and appetite sensation is registered three times daily before the main meals.

ELIGIBILITY:
Inclusion Criteria:

* 18-40y
* BMI 22-28
* healthy

Exclusion Criteria:

* smoking
* medication
* excess PA

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2009-03; Primary Completion 2009-07 (Actual); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Fat and energy digestibility | mean over period

SECONDARY OUTCOMES:
appetite | three times daily
gastrointestinal distress | continously
lipid profile | end of each period
glucose and insulin | end of each period
fecal output and transit time | mean of each period

CONTACTS AND LOCATIONS:
Overall Officials: Arne Astrup, PhD, Dr med, Principal Investigator — University of Copenhagen
Locations (1):
- University of Copenhagen, Department og Human Nutrition, Frederiksberg C, Denmark

REFERENCES:
- [Derived] Kristensen M, Jensen MG, Aarestrup J, Petersen KE, Sondergaard L, Mikkelsen MS, Astrup A. Flaxseed dietary fibers lower cholesterol and increase fecal fat excretion, but magnitude of effect depend on food type. Nutr Metab (Lond). 2012 Feb 3;9:8. doi: 10.1186/1743-7075-9-8. PMID 22305169